CLINICAL TRIAL: NCT03920072
Title: A Phase 3b Open-label Study of the Anti-FGF23 Antibody, Burosumab (KRN23) in Adult Patients With X-linked Hypophosphatemia (XLH)
Brief Title: Study of the Anti-FGF23 Antibody, Burosumab, in Adults With XLH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUR02
Record Dates: First submitted 2018-10-29; First posted 2019-04-18 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: X-linked Hypophosphatemia
Keywords: Crysvita; Burosumab; X-linked Hypophosphatemia (XLH); PHEX Gene Mutation; PHEXdb
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Intervention Model Description: Open-label, international, multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (Other): All subjects will be administered subcutaneously burosumab every 4 weeks at the dosage defined in study UX023-CL303 or UX023-CL304 until December 2021 or when the drug becomes commercially available.
  Interventions: Drug: Burosumab

INTERVENTIONS:
Drug: Burosumab — Burosumab is a sterile, clear, colourless and preservative free solution supplied in single-use 5ml vials containing 1mL of burosumab at a concentration of 30mg/mL
  Other Names: KRN23; Crysvita

SUMMARY:
This is phase 3b open-label, international, multicenter study to continue to monitor the long-term safety and efficacy of burosumab in adult patients with XLH that participated in previous clinical trials with burosumab (UX023-CL303 / UX023-CL304).

DETAILED DESCRIPTION:
XLH is a rare, genetic disorder that is serious, chronically debilitating and represents an unmet medical need. XLH is the most common inherited form of rickets and the most common inherited defect in renal tubular phosphate transport. XLH is transmitted as an X-linked dominant disorder. Mutations resulting in the loss of function of PHEX form the genetic basis for XLH. More than 300 different PHEX gene mutations have been identified in patients with XLH (PHEXdb); however, few definitive correlations have been observed between specific mutations and phenotypic severity.

Patients with XLH have hypophosphatemia due to excessive serum FGF23 levels. FGF23 reduces serum phosphorus levels by two distinct mechanisms of action. The primary mechanism is to inhibit phosphate reabsorption in the proximal tubule of the kidney. The secondary mechanism is to decrease phosphate absorption by the small intestine through the inhibition of 1,25(OH)2D production in the kidney.

Burosumab has the potential to block or reduce FGF23 action and improve phosphate homeostasis in XLH patients. Burosumab binds the amino-terminal domain of FGF23 that interacts with the FGF-binding portion of the combination FGFR1/Klotho receptor, preventing FGF23 from binding to and signaling from its receptor. Both intact and fragmented FGF23 polypeptides are immunoprecipitated with burosumab. By inhibiting FGF23, burosumab restores tubular reabsorption of phosphate (as measured by the ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate [TmP/GFR]) from the kidney and increases the production of 1,25(OH)2D that also enhances intestinal absorption of phosphate. The dual action on kidney reabsorption and intestinal absorption improves serum phosphorus levels, which is expected to improve bone mineralization and reduce the diverse bone and non-bone manifestations associated with hypophosphatemia in XLH patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures.
2. Subjects who participated in Study UX023-CL303 or UX023-CL304. Any subjects that did not complete Study UX023-CL303 or UX023-CL304 may be included on a case-by-case basis. Subjects' enrolment is not dependent on any response to Primary or Secondary endpoints in studies UX023-CL303 or UX023-CL304.
3. Willing to provide access to prior medical records for the collection of historical growth, biochemical and radiographic data, and disease history.
4. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments.
5. Females of child-bearing potential must have a negative urine pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not to be of child-bearing potential include those who have been in menopause for at least two years prior to Screening, or have had tubal ligation at least one year prior to Screening, or have had a total hysterectomy or bilateral salpingo-oophorectomy. If sexually active, male and female subjects must be willing to use one highly effective method of contraception for the duration of the study.

Exclusion Criteria:

1. Hypocalcemia or hypercalcemia, defined as serum calcium levels outside the age-adjusted normal limits and deemed as clinically significant in the opinion of the investigator.
2. Presence of a concurrent disease or condition that would interfere with study participation or affect safety in the opinion of the investigator or Sponsor.
3. Use of any investigational product other than burosumab or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
4. Subjects with major protocol deviations in Study UX023-CL303 or UX023-CL304 which in the view of the investigator places the subject at high risk of poor treatment compliance or of not completing the study.
5. Subjects who discontinued treatment from Study UX023-CL303 or UX023-CL304 due to either a grade ≥3 treatment-related hypersensitivity reaction or a burosumab-related hypersensitivity reaction reported as a SAE.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving mean serum phosphorus levels above the LLN (2.5mg/dL[0.81mmol/L]), as averaged across dose cycles between baseline and their last administered dose. | Serum phosphorous levels will be monitored from Screening and every 12 weeks until the end of the study, at approximately 144 weeks.
  To establish the effect of burosumab treatment on maintaining serum phosphorus levels to within normal range in adults with XLH.

SECONDARY OUTCOMES:
Effect of burosumab on pre-existing pseudofracture healing will be monitored by centrally read targeted X-Ray | Targetted X-Rays at ongoing fracture sites will be taken at the End of Study Visit, approximately week 144.
  Targeted radiography at locations pre-determined by the skeletal survey performed during UX023-CL303 or UX023-CL304 will be taken to monitor healing of pseudofractures and/or fractures.
Effect of burosumab on patients walking ability measured using the 6 Minute Walk Test. | The 6MWT will be measured at Baseline and then every 12 weeks for the first 48 weeks and then every 24 weeks for up to 144 weeks
  Patient's motor function by sustained walking will be evaluated using the 6 Minute Walk Test. (6MWT). The percent predicted values for the 6MWT will be calculated using published normative data based on age, gender and height.
Effect of burosumab on Patient mobility assessed using the Timed Up and Go Test (TUG). | The TUG Test will be assessed at Baseline and then every 12 weeks for the first 48 weeks and then every 24 weeks for up to 144 weeks
  The TUG assesses transitions during ambulatory activity incorporating strength, agility and dynamic balance assessments. The TUG score will be reported as the time (in seconds) that a subject takes to rise from a chair, walk three meters (approximately 10 feet), turn around, walk back to the chair and sit down.
Effect of burosumab on stiffness and physical function will be assessed using WOMAC. | The WOMAC questionnaire will be administered at Baseline and then every 12 weeks for 48 weeks and every 12 weeks for up to 48 weeks and then every 24 weeks for up to 96 weeks
  The patient's impression of their stiffness and physical function will be assessed by administering the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire- a 24 item patient reported questionnaire. The WOMAC will be administered in a 5-point Likert-scale format using descriptors of none, mild, moderate, severe and extreme corresponding to an ordinal scale of 0 to 4. Higher scores on the WOMAC indicate worse stiffness and functional limitations.
Effect of burosumab on patient's pain severity and the impact of pain on functioning will be assessed using the Short-form Brief Pain Inventory questionnaire. | The BPI will be administered at Baseline and then every 12 weeks for 48 weeks and then every 24 weeks for up to 144 weeks
  The patient's recall of pain over a 24 hour period will be captured by administering the short form of the Brief Pain Inventory (BPI) questionnaire. The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others and sleep).
Effect of burosumab on patient's fatigue and the interference of fatigue on daily life over a 24 hour period. | The BFI will be administered at Baseline and then every 12 weeks for up to 48 weeks and then every 12 weeks for up to 144 weeks
  The patient's recall of fatigue will be captured by administering the Brief Fatigue Inventory (BFI) questionnaire. The BFI is a self-reported questionnaire consisting of nine items related to fatigue that are rated on a 0 to 10 numerical rating scale with a recall period of 24 hours. Two dimensions are measured: fatigue and the interference of fatigue on daily life. The change from baseline to post-baseline visits will be assessed.
Effect of burosumab on bone metabolism and phosphate homeostasis using urinary phosphorus as PD marker. | Pharmacodynamic analysis will be conducted at Baseline and every 12 weeks for up to 88 weeks
  Pharmacodynamic assessment.
Effect of burosumab on enthesopathy will be monitored by centrally read targeted X-Ray. | Lateral foot views (bilateral) will be obtained at screening and at End of Study, approximately week 88.
  Lateral foot views (bilateral) will be obtained in all subjects at Screening (as part of skeletal survey) and at End of Study (EOS). Size of enthesopathy spurs at both the superior and inferior calcaneus will be measured in two dimensions.
Effect of burosumab on bone metabolism and phosphate homeostasis using Serum Phosphorus as PD marker. | Pharmacodynamic analysis will be conducted at Baseline and every 12 weeks for up to 88 weeks.
  Pharmacodynamic assessment.
Effect of burosumab on bone metabolism and phosphate homeostasis using serum 1, 25(OH)2D as PD marker. | Pharmacodynamic analysis will be conducted at Baseline and every 12 weeks for up to 88 weeks.
  Pharmacodynamic assessment.
Effect of Burosumab on phosphate reabsorption as measured by the ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtrate [TmP/GFR]. | Pharmacodynamic analysis will be conducted at Baseline and every 12 weeks for up to 88 weeks.
  Pharmacodynamic assessment.
Effect of burosumab on health related quality of life as measured by SF-36v2 | The SF-36v2 will be administered at Baseline and then every 12 weeks for 48 weeks and then every 24 weeks for up to 144 weeks
  Patients will answer questions around their physical functioning, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kamenicky, Principal Investigator — CHU de Bicêtre
Locations (10):
- France (3):
  - CHU de Bicetre, Le Kremlin-Bicêtre
  - Hopital Lariboisiere, Paris
  - Hopital Cochin, Paris
- St. Vincent's University Hospital, Dublin, Ireland
- Azienda ospedaliera universitaria Careggi, Florence, Italy
- United Kingdom (5):
  - Western General Hospital, Edinburgh
  - National Hospital for Neurology and Neurosurgery-University College London Hospitals NHS Foundation Trust, London
  - Nuffield Orthopaedic Centre - Oxford University Hospitals Nhs Trust, Oxford
  - Northen General Hospital, Sheffield
  - Royal National Orthopaedic Hospital NHS Trust, Stanmore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamenicky P, Briot K, Brandi ML, Cohen-Solal M, Crowley RK, Keen R, Kolta S, Lachmann RH, Lecoq AL, Ralston SH, Walsh JS, Rylands AJ, Williams A, Sun W, Nixon A, Nixon M, Javaid MK. Benefit of burosumab in adults with X-linked hypophosphataemia (XLH) is maintained with long-term treatment. RMD Open. 2023 Feb;9(1):e002676. doi: 10.1136/rmdopen-2022-002676. PMID 36854566